CLINICAL TRIAL: NCT02530723
Title: The Effects of Low-intensity Power Training on Strength, Power, and Functional Outcomes in Older, Community-dwelling Women.
Brief Title: Functional Changes and Power Training in Older Women.
Acronym: F-POW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Konstantina Katsoulis, Konstantina Katsoulis, University of Toronto
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 27773
Record Dates: First submitted 2015-08-17; First posted 2015-08-21 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Sarcopenia; Muscle Weakness
Keywords: power training; high-speed training; high-velocity training; function; older adults; older women
MeSH Terms: conditions — Sarcopenia; Muscle Weakness | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: With 3 groups and a wait-control group, our general design will include 4 (group) x 2 (baseline and post-study) and 4 (group) x 3 (baseline, midpoint, and post-study) analyses. We may also conduct one-way ANOVA analyses as problems with normality in the data are apparent.
Who Masked: Outcomes Assessor
Masking Description: Functional testers are masked to what group the participants are in (control, Exercise Group I, II, or III). All testers are masked during baseline testing.
Oversight: Data Monitoring Committee: No

ARMS (4):
- Once a week (Experimental): Group 1 will be invited to perform resistance training exercise 1 day/week. After a 2-week familiarization phase, participants will engage in power training (40% of 1-repetition maximum) for 12 weeks. Instructions include telling participants to lift the weight concentrically 'as fast as possible', with a lowering phase (eccentric) of 2-3 seconds. Participants will perform 3 x 12-14 repetitions per exercise per session. Primarily lower body equipment will be used, including leg press, knee extension/flexion, hip extension/flexion, and calf-raises.
  Interventions: Other: power training
- Twice a week (Experimental): Group 2 will be invited to perform resistance training exercise 2 days/week. After a 2-week familiarization phase, participants will engage in power training (40% of 1-repetition maximum) for 12 weeks. Instructions include telling participants to lift the weight concentrically 'as fast as possible', with a lowering phase (eccentric) of 2-3 seconds. Participants will perform 3 x 12-14 repetitions per exercise per session. Primarily lower body equipment will be used, including leg press, knee extension/flexion, hip extension/flexion, and calf-raises.
  Interventions: Other: power training
- Thrice a week (Experimental): Group 3 will be invited to perform resistance training exercise 3 days/week. After a 2-week familiarization phase, participants will engage in power training (40% of 1-repetition maximum) for 12 weeks. Instructions include telling participants to lift the weight concentrically 'as fast as possible', with a lowering phase (eccentric) of 2-3 seconds. Participants will perform 3 x 12-14 repetitions per exercise per session. Primarily lower body equipment will be used, including leg press, knee extension/flexion, hip extension/flexion, and calf-raises.
  Interventions: Other: power training
- wait-control (No Intervention): Participants in this group will serve as controls prior to participating in power training in 1 of the above treatment groups. The control period will last as long as the exercise period, or 3 months. Controls will participate in the same testing time points as the exercisers (baseline, midpoint, and post-intervention).

INTERVENTIONS:
Other: power training — Resistance training machines with CAM devices will be used for training.
  Other Names: resistance training; high-speed training; high-velocity training
  Arms: Once a week; Thrice a week; Twice a week

SUMMARY:
Extending quality of life and attenuating functional decline is paramount in older adults. This study investigates the effects of low-intensity power-training in older women and its effects on functional outcomes.

DETAILED DESCRIPTION:
Resistance training has gained popularity in aging interventions since it is effective in countering the loss of muscle mass and strength with senescence. Traditionally, strength training (ST) protocols for the elderly have involved relatively heavy loads (70-80% of maximum force) with the focus being on increasing strength. There is some evidence of increased function after strength training albeit with inconsistent reports in the literature. More recently, several studies have designed resistance training programs that aim to increase power rather than strength, since findings indicate that measures of power are better predictors of physical function than measures of strength. In other words, improving power may be more beneficial to the elderly who are susceptible to functional limitations, mobility disability, and dependency. Since it is difficult to produce a great deal of power with increasing intensities, and lifting heavy loads may not be relevant to everyday functioning in the elderly, studies have investigated training for improvements in power rather than the traditional improvements in strength.

The effects of power training (PT) versus ST on functional outcomes in older adults have varied, with some studies showing enhanced improvements in function, and others showing no difference in function compared to regular ST or compared to other interventions such as walking. Discrepancies might be the result of the variety of functional tests used, mode of training, variable frequency of sessions per week, differences in study length, and adults of varying functional status. It has been suggested that perhaps the standard 3-sessions-per-week frequency may not be optimal for the elderly. A previous investigation demonstrated that the effects from PT at 40% of the 1-repetition maximum (1RM: the highest amount that can be lifted once) in older adults was comparable to the effects from ST at 80% 1RM with improvements being similar between the two modes despite the lower daily ratings of perceived exertion (RPE) reported with PT (PT: RPE for leg press (12.2) and knee extension (14.6) vs ST: RPE for leg press (15.1) and knee extension (17)). Therefore, an 'easier' exercise training experience did not result in sacrifices in gains of strength and power. In theory, these factors (lighter loads, lower perceived exertions, similar strength and power gains) could affect adherence to exercise during and after a research-related exercise intervention has been completed and thus are important considerations in the design of a training program.

The purpose of this research is to investigate the effects of low-intensity (40% 1RM) PT on functional outcomes in older women.

ELIGIBILITY:
Inclusion Criteria:

* females, 65 years of age
* agree to the study protocol
* give informed-consent to the proposed research study

Exclusion Criteria:

* existing acute illness/disease (last six months)
* diagnosed with myopathies
* currently prescribed cardiovascular medications or drugs that may affect muscle mass and/or their response to exercise (thyroid medications, sedatives, beta blockers, some statins)
* are diabetic
* have uncontrolled hypertension
* have been advised against participating in exercise by their doctor

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-16 (Actual)

PRIMARY OUTCOMES:
Change in Stair-climb power | baseline, 6 weeks, 12 weeks
  The time needed to ascend a flight of stairs, converted to power (using body-weight and stair height)

SECONDARY OUTCOMES:
Change in 400-meter walk test | baseline, 6 weeks, 12 weeks
  The time needed to walk 400 meters (back and forth along a 20 meter course)
Change in Short Physical Performance Battery | baseline, 6 weeks, 12 weeks
  A short test of balance, walking, and chair stand ability
Change in 30-second chair stand test | baseline, 6 weeks, 12 weeks
  The number of chair stands possible in 30 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Catherine E Amara, Ph.D, Study Director — University of Toronto; Faculty of Kinesiology and Physical Education
Locations (1):
- Athletic Centre; 55 Harbord Street, Toronto, Ontario, Canada

REFERENCES:
- [Background] Fiatarone MA, O'Neill EF, Ryan ND, Clements KM, Solares GR, Nelson ME, Roberts SB, Kehayias JJ, Lipsitz LA, Evans WJ. Exercise training and nutritional supplementation for physical frailty in very elderly people. N Engl J Med. 1994 Jun 23;330(25):1769-75. doi: 10.1056/NEJM199406233302501. PMID 8190152
- [Background] Hartman MJ, Fields DA, Byrne NM, Hunter GR. Resistance training improves metabolic economy during functional tasks in older adults. J Strength Cond Res. 2007 Feb;21(1):91-5. doi: 10.1519/00124278-200702000-00017. PMID 17313273
- [Background] Hanson ED, Srivatsan SR, Agrawal S, Menon KS, Delmonico MJ, Wang MQ, Hurley BF. Effects of strength training on physical function: influence of power, strength, and body composition. J Strength Cond Res. 2009 Dec;23(9):2627-37. doi: 10.1519/JSC.0b013e3181b2297b. PMID 19910811
- [Background] Pojednic RM, Clark DJ, Patten C, Reid K, Phillips EM, Fielding RA. The specific contributions of force and velocity to muscle power in older adults. Exp Gerontol. 2012 Aug;47(8):608-13. doi: 10.1016/j.exger.2012.05.010. Epub 2012 May 22. PMID 22626972
- [Background] Sayers SP, Guralnik JM, Thombs LA, Fielding RA. Effect of leg muscle contraction velocity on functional performance in older men and women. J Am Geriatr Soc. 2005 Mar;53(3):467-71. doi: 10.1111/j.1532-5415.2005.53166.x. PMID 15743291
- [Background] Miszko TA, Cress ME, Slade JM, Covey CJ, Agrawal SK, Doerr CE. Effect of strength and power training on physical function in community-dwelling older adults. J Gerontol A Biol Sci Med Sci. 2003 Feb;58(2):171-5. doi: 10.1093/gerona/58.2.m171. PMID 12586856
- [Background] Sayers SP, Gibson K. Effects of high-speed power training on muscle performance and braking speed in older adults. J Aging Res. 2012;2012:426278. doi: 10.1155/2012/426278. Epub 2012 Feb 28. PMID 22500229
- [Background] Henwood TR, Riek S, Taaffe DR. Strength versus muscle power-specific resistance training in community-dwelling older adults. J Gerontol A Biol Sci Med Sci. 2008 Jan;63(1):83-91. doi: 10.1093/gerona/63.1.83. PMID 18245765
- [Background] Drey M, Zech A, Freiberger E, Bertsch T, Uter W, Sieber CC, Pfeifer K, Bauer JM. Effects of strength training versus power training on physical performance in prefrail community-dwelling older adults. Gerontology. 2012;58(3):197-204. doi: 10.1159/000332207. Epub 2011 Nov 3. PMID 22056537
- [Background] Earles DR, Judge JO, Gunnarsson OT. Velocity training induces power-specific adaptations in highly functioning older adults. Arch Phys Med Rehabil. 2001 Jul;82(7):872-8. doi: 10.1053/apmr.2001.23838. PMID 11441371
- [Background] Bamman MM, Hill VJ, Adams GR, Haddad F, Wetzstein CJ, Gower BA, Ahmed A, Hunter GR. Gender differences in resistance-training-induced myofiber hypertrophy among older adults. J Gerontol A Biol Sci Med Sci. 2003 Feb;58(2):108-16. doi: 10.1093/gerona/58.2.b108. PMID 12586847
- [Background] Hunter GR, Wetzstein CJ, McLafferty CL Jr, Zuckerman PA, Landers KA, Bamman MM. High-resistance versus variable-resistance training in older adults. Med Sci Sports Exerc. 2001 Oct;33(10):1759-64. doi: 10.1097/00005768-200110000-00022. PMID 11581563
- [Derived] Katsoulis K, Amara CE. The Effects of Power Training Frequency on Muscle Power and Functional Performance in Older Women: A Randomized Controlled Trial. J Strength Cond Res. 2023 Nov 1;37(11):2289-2297. doi: 10.1519/JSC.0000000000004527. Epub 2023 Jun 19. PMID 37335760